CLINICAL TRIAL: NCT01156987
Title: Improved Breast Dynamic Contrast Enhanced-magnetic Resonance Imaging (DCE-MRI) With Sweep Imaging With Fourier Transform (SWIFT)
Brief Title: Improved Breast MRI With SWIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009NTLS055; 0907M69461 (Other: IRB, University of Minnesota); 1R21CA139688 (NIH)
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Volunteers (Experimental): Five healthy women will be screened for Magnetic Resonance Imaging (MRI) contraindications, and then undergo contrast injection, and SWIFT acquisition.
  Interventions: Device: Magnetic resonance imaging
- Breast Cancer Patients (Experimental): 40 breast cancer patients who have suspected breast lesion that will be biopsied will be screened for Magnetic Resonance Imaging (MRI) contraindications, and then undergo contrast injection and SWIFT acquisition.
  Interventions: Device: Magnetic resonance imaging

INTERVENTIONS:
Device: Magnetic resonance imaging — Patients and healthy volunteers will be first screened for MRI contraindications. The SWIFT MRI workflow will be performed as follows:
  * an IV line is placed by nurse,
  * patient is placed in the 4 T MRI scanner at CMRR,
  * initial scout images and manual linear shims are adjusted,
  * Pre-contrast SWIFT T1 weighted images and T1 map are obtained,
  * continuous SWIFT acquisition begins immediately before contrast injection,
  * contrast injection,
  * continuous SWIFT acquisition continues for 12 min after contrast,
  * late enhancement images may also be obtained.
    10 and 30 patients will be scanned in the first and second year, respectively. Thresholds will be set for prospective analysis. SWIFT-DCE diagnostic performance will be compared to prior FLASH-DCE methods.
  Other Names: SWIFT

SUMMARY:
Today's medical imaging methods have insufficient specificity for reliable differentiation between benign and malignant breast lesions in patients. Pathologic evaluation is currently the only way to obtain a definitive diagnosis. This research will use a novel method of magnetic resonance imaging (MRI), Sweep Imaging with Fourier Transform (SWIFT), at a very high magnetic field (4 Tesla) to distinguish malignant from benign breast lesions. This research will reveal whether the SWIFT sequence bears new capabilities in medical imaging for breast cancer diagnosis.

DETAILED DESCRIPTION:
Patients will be asked to come to the Center for Magnetic Resonance Research (CMRR) at the University of Minnesota. Researchers will interview the patient and describe procedures and risks. An intravenous (IV) line will be placed in an upper extremity for infusing magnetic resonance imaging (MRI) contrast dye. Baseline MRI scans will be done. These MRI measurements will be compared with clinical, radiological and pathological findings (the gold standard).

Follow-up contact will occur within one year after the MRI to determine whether a pathology report is available.

ELIGIBILITY:
Inclusion Criteria:

* Women with a clinically or mammographically identified suspicious breast mass that is likely to be biopsied or surgically removed.

Exclusion Criteria:

* Pregnancy
* Ferromagnetic implants
* History of shotgun wounds and shrapnel
* Obesity (>250 pounds)
* Cardiac pacemaker
* Incompatible implanted medical device
* Severe claustrophobia
* Major surgeries with potential of ferromagnetic implants
* Severe asthma and allergies
* i-STAT system, a handheld blood analyzer (I-STAT) creatinine test, estimated glomerular filtration rate (GFR) <30
* Metallic object (greater than 2 cm in length) in the breast
* Metallic ink tatoo within 20 cm of the breast (approximately 8 inches)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Corum, Ph.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Center for Magnetic Resonance Research, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Corum CA, Idiyatullin D, Snyder CJ, Garwood M. Gap cycling for SWIFT. Magn Reson Med. 2015 Feb;73(2):677-82. doi: 10.1002/mrm.25141. Epub 2014 Feb 24. PMID 24604286
- [Background] Idiyatullin D, Corum C, Park JY, Garwood M. Fast and quiet MRI using a swept radiofrequency. J Magn Reson. 2006 Aug;181(2):342-9. doi: 10.1016/j.jmr.2006.05.014. Epub 2006 Jun 19. PMID 16782371
- [Result] Nelson MT, Benson JC, Prescott T, Corum CA, Snyder A, Garwood M. Breast MRI using SWeep Imaging with Fourier Transform (SWIFT). Eur J Radiol. 2012 Sep;81 Suppl 1(0 1):S109. doi: 10.1016/S0720-048X(12)70044-X. No abstract available. PMID 23083549
- [Result] Corum CA, Benson JC, Idiyatullin D, Snyder AL, Snyder CJ, Hutter D, Everson LI, Eberly LE, Nelson MT, Garwood M. High-spatial- and high-temporal-resolution dynamic contrast-enhanced MR breast imaging with sweep imaging with Fourier transformation: a pilot study. Radiology. 2015 Feb;274(2):540-7. doi: 10.1148/radiol.14131273. Epub 2014 Sep 22. PMID 25247405

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 were consented to enroll to start study with 23 breast cancer subjects and 8 healthy controls being able to complete the portion of the MRI study needed for analysis.
Groups:
- Healthy Volunteers: Healthy women will be screened for Magnetic Resonance Imaging (MRI) contraindications, and then undergo contrast injection, and SWIFT acquisition.
  Magnetic resonance imaging: Patients and healthy volunteers will be first screened for MRI contraindications. The SWIFT MRI workflow will be performed as follows:
  * an IV line is placed by nurse,
  * patient is placed in the 4 T MRI scanner at CMRR,
  * initial scout images and manual linear shims are adjusted,
  * Pre-contrast SWIFT T1 weighted images and T1 map are obtained,
  * continuous SWIFT acquisition begins immediately before contrast injection,
  * contrast injection,
  * continuous SWIFT acquisition continues for 12 min after contrast,
  * late enhancement images may also be obtained.
    10 and 30 patients will be scanned in the first and second year, respectively. Thresholds will be set for prospective analysis. SWIFT-DCE diagnostic performance will be compared to prior FLASH-DCE methods.
- Breast Cancer Patients: Breast cancer patients who have suspected breast lesion that will be biopsied will be screened for Magnetic Resonance Imaging (MRI) contraindications, and then undergo contrast injection and SWIFT acquisition.
  Magnetic resonance imaging: Patients and healthy volunteers will be first screened for MRI contraindications. The SWIFT MRI workflow will be performed as follows:
  * an IV line is placed by nurse,
  * patient is placed in the 4 T MRI scanner at CMRR,
  * initial scout images and manual linear shims are adjusted,
  * Pre-contrast SWIFT T1 weighted images and T1 map are obtained,
  * continuous SWIFT acquisition begins immediately before contrast injection,
  * contrast injection,
  * continuous SWIFT acquisition continues for 12 min after contrast,
  * late enhancement images may also be obtained. 10 and 30 patients will be scanned in the first and second year, respectively. Thresholds will be set for prospective analysis. SWIFT-DCE diagnostic performance will be compar
Period: Overall Study
Arm/Group | Healthy Volunteers | Breast Cancer Patients
Started | 8 | 23
Completed | 8 | 12
Not Completed | 0 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Breast Cancer Patients | Total
Number analyzed (Participants) | 8 | 23 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 23 | 31
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 23 | 31
  Male | 0 | 0 | 0
Lesion measurements [Number; unit: participants] | 8 | 23 | 31

OUTCOME MEASURES:

1. Primary Outcome: Lesions
Description: Number of lesions detected
Time Frame: at time of read by two radiologiests, compared to biopsy within 7 days.
Measure: Number; unit: lesions
Arm/Group | Healthy Volunteers | Breast Cancer Patients
Number analyzed (Participants) | 8 | 23
lesions | 0 | 12

ADVERSE EVENTS:
Arm/Group | Healthy Volunteers | Breast Cancer Patients
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/23
Other Adverse Events (participants affected / at risk) | 0/8 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No